CLINICAL TRIAL: NCT05248789
Title: Efficacy and Safety Study of Oncolytic Virus (OH2) Intratumoral Injection in Locally Advanced or Metastatic Bladder Cancer a Phase Ⅱ Clinical Trial
Brief Title: OH2 Oncolytic Viral Therapy in Advanced Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategy adjustment
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-OH2-017
Record Dates: First submitted 2022-01-27; First posted 2022-02-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-08

CONDITIONS: Advanced Bladder Carcinoma
Keywords: Oncolytic Virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OH2 (Experimental): OH2 dosage: 1x10e7 CCID50/mL Administration：intratumoral injection Frequency：once two weeks
  Interventions: Biological: OH2 injection

INTERVENTIONS:
Biological: OH2 injection — OH2: Oncolytic Type 2 Herpes Simplex Virus

SUMMARY:
This Ⅱ study evaluates the safety and efficacy of intratumoral injection of OH2 in locally advanced or metastatic bladder cancer.

OH2 is an oncolytic virus developed upon genetic modifications of the herpes simplex virus type 2 strain HG52, allowing the virus to selectively replicate in tumors. Meanwhile, the delivery of the gene encoding human granulocyte macrophage colony-stimulating factor (GM-CSF) may induce a more potent antitumor immune response.

DETAILED DESCRIPTION:
This is a phase Ⅱ study evaluating the efficacy and safety of OH2 in locally advanced or metastatic bladder cancer.

BH-OH2-017 is a single-arm,multicenter clinical trial. The OH2 injection will be delivered once two weeks. In the maintenance treatment period, OH2(1x10e7 CCID50/mL) will be delivered once a month.

Adverse events (AEs) are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).

Radiographic imaging studies are performed using computed tomography or magnetic resonance imaging. Measurement of cutaneous or subcutaneous lesions are conducted with calipers. Evaluation of response are performed by the investigators using both the RECIST version 1.1 and the iRECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to sign informed consent, willing to follow the study procedures.
2. Age 18 ~ 75 years old (including boundary value), male or female.
3. ECOG 0-1.
4. Histologically or cytologically confirmed advanced bladder cancer，relapsed and metastasized after radiotherapy or immunotherapy.
5. Life expectancy >12 weeks.
6. Agree to provide last surgical specimens (including paraffin blocks, paraffin embedded sections, etc.).
7. At least 6 weeks after previous anti-tumor treatment (radiotherapy, chemotherapy and immunotherapy) and the first administration of this trial.
8. Appropriate organ function and hematopoietic function: neutrophil count (neut ≥ 1.5 × 109/L； White blood cell count (WBC) ≥ 3.0 × 109/L； Platelet count ≥ 100 × 109/L； Hemoglobin ≥ 90g / L; Serum creatinine ≤ 1.5 times the upper limit of normal value (ULN); AST and alt ≤ 2.5 times ULN; Serum total bilirubin ≤ 1.5 times ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 times ULN (except for patients undergoing anticoagulant therapy).
9. Agree to take effective contraceptive measures during treatment and at least 180 days after the last treatment.

Exclusion Criteria:

1. The primary tumor was upper urinary tract and ureteral urothelial carcinoma.
2. Malignant tumors other than bladder urothelial carcinoma within 5 years before enrollment.

   except:

   ①Prostate cancer with local low risk (stage ≤ T2b, Gleason score ≤ 7, PSA ≤ 20ng / ml, no recurrence after treatment (judged by reviewing PSA level)).

   ②Low risk prostate cancer (stage T1 / T2a, Gleason score ≤ 7, and PSA ≤ 10NG / ml, in the observed but untreated stage.

   ③For malignant tumors that meet other inclusion criteria but have a very low risk of metastasis or death, after standard treatment, recheck the patients whose imaging and disease-specific tumor markers show no recurrence or metastasis, such as fully treated cervical cancer in situ, basal or squamous cell skin cancer; Ductal carcinoma in situ after treatment and operation.
3. Active autoimmune diseases and need systemic treatment in the past two years (i.e. long-term use of corticosteroids or immunosuppressive drugs). Alternative therapies (such as thyroxine, insulin or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) are excluded.
4. Expected to have major surgery during the study period or had major surgery within 4 weeks before administration.
5. Received other vaccines within 30 days before the first administration (including new crown vaccine)
6. Any immune related toxicity caused by previous cancer treatment did not return to ≤ grade 1 (except for grade 2 endocrine system diseases receiving stable dose hormone replacement therapy), and / or any other toxicity related to previous anti-cancer treatment (except immune related toxicity) did not return to ≤ grade 2, except hair loss.
7. Human immunodeficiency virus (HIV) seropositive or history of HIV infection or other acquired immunodeficiency diseases.
8. Long-term use of antiviral drugs, including hepatitis B (HBsAg positive and HBV DNA equal to 2000 IU/ml at the same time, and excluding hepatitis or other causes of hepatitis), hepatitis C (at the same time to meet the anti HCV antibody positive, and HCV-RNA fruit is greater than the lower limit).
9. Uncontrolled systemic diseases, such as cardiovascular and cerebrovascular diseases and diabetes.
10. History of organ transplantation or stem cell transplantation.
11. Cardiac insufficiency (patients classified as III-IV according to NY-HA of New York Heart Association).
12. Lung disease (such as shortness of breath during rest or slight activity or oxygen supplement for any reason).
13. Other basic diseases which would interfere with the diagnosis of the disease, or might potentially cause serious complications
14. Other serious infections before administration
15. Alcohol addicts or history of drug abuse.
16. History of neurological or mental disorders, such as epilepsy, dementia, poor compliance, or peripheral nervous system disorders.
17. Pregnancy or lactation, or expected pregnancy or childbirth during the trial period.
18. Allergic to study drug or have a history of allergic reaction to the main and auxiliary materials of any dosage form in the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  The assessment result is the number and proportion of subjects with complete response + partial response.

SECONDARY OUTCOMES:
Disease Control Rate | 2 years
  The assessment result is the number and proportion of subjects with complete response + partial response + stable disease.
Progression-Free Survival | 2 years
  Time after OH2 administration to clinical and radiographic disease progression will be evaluated.
Overall Survival | 5 years
  The overall survival for each patient receiving OH2 will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China